CLINICAL TRIAL: NCT04961489
Title: Impact of Measures Taken to Contain COVID-19 on Hospital Surgical Care Services and Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020/2706
Record Dates: First submitted 2021-07-12; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Surgery
Keywords: Covid-19 pandemic; emergency; cancer; elective surgery; postponement
MeSH Terms: conditions — COVID-19; Emergencies; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to look at the impact on patient outcomes arising from measures implemented during the COVID-19 pandemic. The information and knowledge from this study will be useful for the management and allocation of hospital resources and patients in tne event of a disease outbreak.

ELIGIBILITY:
Inclusion Criteria:

* This study involves the extraction of patient records from the enterprise dataware house. As such, we do not stipulate the age limits.
* Patients who had the following surgeries during over the period of 1 Jan 2017 to 31 December 2020
* From the identified surgical procedure type or the following cancer-related procedures:

  1. Breast
  2. Colon
  3. Liver
  4. Rectum
* Selected non-cancer surgeries:

  1. Abdominal Wall
  2. Gallbladder
* Patients from SGH and its related institute NCC
* Only local Singapore Citizens

Exclusion Criteria:

* No exclusion criteria

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study seeks to assess the effect of the measures taken to contain COVID 19 on patients who need surgical services measured by patient outcomes, such as, length of hospital stay (LOS), ICU stay, APACHE score, and stage of cancer at surgery.
Sampling Method: Probability Sample
Enrollment: 11000 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Analysis of patients according to type of surgical procedures, medical condition and dates of surgical treatment retrospectively. | 1 Jan - 31 Dec 2017, 1 Jan - 31 Dec 2018, 1 Jan - 31 Dec 2019, 1 Jan - 31 Dec 2020
  These patients are classified according to the institution, type of surgical procedures, the medical condition and the dates of surgical treatment. The study will be compared across four time periods.
Comparing surgical indices for high volume cancer and non-cancer diagnoses | 1 Jan 2020 - 31 Dec 2020
  The study focus on surgical indices for selected high-volume cancer and non-cancer diagnoses over the period 1st January2020 to 31 December 2020 and compare them with similar indices across the same period of time in the preceding 3 years in particular, for the following surgical procedures:
  1. Surgeries for the following cancer diagnoses:
     1. breast cancer, [XIV- N60, no malignancy], [Malignant, IINeoplasms- C50], colorectal cancer, [C18, 19, 20],
     2. hepatocellular carcinoma, [C22]
  2. Selected non-cancer surgeries:
     1. Cholecystectomy
     2. Abdominal hernia repair

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Chow, MD, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - National Cancer Center Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazingi D, Navarro S, Bobel MC, Dube A, Mbanje C, Lavy C. Exploring the Impact of COVID-19 on Progress Towards Achieving Global Surgery Goals. World J Surg. 2020 Aug;44(8):2451-2457. doi: 10.1007/s00268-020-05627-7. PMID 32488665
- [Background] Al-Jabir A, Kerwan A, Nicola M, Alsafi Z, Khan M, Sohrabi C, O'Neill N, Iosifidis C, Griffin M, Mathew G, Agha R. Impact of the Coronavirus (COVID-19) pandemic on surgical practice - Part 2 (surgical prioritisation). Int J Surg. 2020 Jul;79:233-248. doi: 10.1016/j.ijsu.2020.05.002. Epub 2020 May 12. PMID 32413502
- See also: A Comparison of Statistical Modeling Strategies for Analyzing Length of Stay after CABG Surgery. Health Services and Outcomes Research Methodology — https://link.springer.com/article/10.1023%2FA%3A1024260023851